CLINICAL TRIAL: NCT02205112
Title: A Multi-center, Randomized, Double-Blind, Parallel Comparative, Phase III Study to Evaluate the Efficacy and Safety of Intravenous Infusion of Nemonoxacin Versus Levofloxain in Treating Adult Patients With CAP
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of Intravenous Infusion of Nemonoxacin in Treating CAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-873870-C-6
Record Dates: First submitted 2014-07-27; First posted 2014-07-31 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Community-acquired Pneumonia
Keywords: intravenous nemonoxacin; community-acquired pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — nemonoxacin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nemonoxacin 500 mg (Experimental): Nemonoxacin 500mg/250mL, intravenous administration, once daily for 7~14 days
  Interventions: Drug: Nemonoxacin
- Levofloxacin 500mg (Active Comparator): Levofloxacin: 500mg/100mL, intravenous administration, once daily for 7~14 days
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Nemonoxacin
  Arms: Nemonoxacin 500 mg
Drug: Levofloxacin
  Arms: Levofloxacin 500mg

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of intravenous nemonoxacin compared with intravenous moxifloxacin in adult patients with community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
Community-acquired Pneumonia (CAP) remains a leading cause of death in both developing and developed countries. In the choice of antibacterial agents used to treat CAP, fluoroquinolones have received considerable attention because of their wide spectrum of bactericidal activity. TG-873870 (Nemonoxacin), a non-fluorinated quinolone (NFQ), is a selective bacterial topoisomerase inhibitor.

This study will evaluate the clinical efficacy, microbiological efficacy and safety of Intravenous nemonoxacin compared with Intravenous levofloxacin in adult patients with community-acquired pneumonia.

Besides, the populationpharmacokinetics (PPK) of nemonoxacin in adult patients with CAP after continuous IV Infusion and the pharmacokinetic (PK)/pharmacodynamic (PD)are to be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 80;
2. Weighs between 40 ~ 100 kg, and BMI ≥ 18 kg/m2;
3. Must have a clinical diagnosis of CAP
4. Chest X-ray and /or CT scan show new or persist/progressive infiltrates
5. Patients with PORT/PSI score II, III or IV.
6. If female, non-lactating and at no risk or pregnancy (post-menopausal or must use adequate birth control)
7. Male must use a reliable form of contraception.
8. Able to receive an intravenous infusion of the drug
9. Able to provide an adequate sputum and blood samples
10. Able to provide written informed consent

Exclusion Criteria:

1. Patients with PORT/PSI score I or VI.
2. Severe CAP is present if a patient needs invasive mechanical ventilation or requires vasopressors.
3. Healthcare-associated pneumonia, hospital-acquired pneumonia, or hospitalized within 14 days before enrollment
4. Virus pneumonia, aspiration pneumonia, ventilator associated pneumonia, or intersstitial lung disease
5. Bronchial bostruction (exclusive of COPD), bronchiectasis, cystic fibrosis, known or suspected pneumocystis pneumonia, known or suspected tuberculosis, primary empyema thoracis, lung abscess, known or suspected lung cancer, or lung disease associated with autoimmune disorders.
6. Medical history of QT prolongation, require the treatment of arrhythmia using class IA or class III drugs, or NYHA functional class >/= III
7. Clinically significant findings on 12-lead ECG, QTc interval>450ms or potassium is < 3.5 mmol/L or lower limit of normal at Screening
8. Immunocompromising illness, such as HIV infection
9. Fatal progressive disease or neurodegenerative diseases that prevent patients from effectively clearing pulmonary secretions
10. Have medical history of seizure, alcohol or drug abuse, suicide tendency, or psychosis that can effect the compliance
11. Have diseases that may affect intravenous infusion.
12. Active hepatitis or decompensated cirrhosis with ascites (Child-Pugh score 10-15/class C);
13. Renal Insufficiency or creatinine >/= 1.1 ULN within 24 hr before first dose
14. ALT or AST >/= 3x ULN, or BUN >/= 30 mg/dL within 24 hr before first dose
15. Neutrophil < 1000 mm3 within 24 hr before first dose
16. Received systemic antibiotics within 72 hr before first dose
17. Received probenecid within 24 hr before first dose or require the treatment with probenecid during study
18. Received quinolones or fluoroquinolones within 14 days before first dose
19. Received any investigational drugs within 30 days before first dose
20. Require the treatment with other systemic antibiotics during study
21. Patients who are being or will be on a long-term medication (over 2 weeks) of steroids (20mg/day)
22. Medical history of hypersensitivity to any quinolone, fluoroquinolone-associated tendinitis and tendon rupture, or myasthenia gravis
23. Current condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the data
24. Participated and received the study medication in previous clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Per subject clinical cure rate | end of treatment and 7 to 14 days after the end of treatment
  The clinical cure rate will be evaluated according to signs and symptoms and changes in the chest X-ray

SECONDARY OUTCOMES:
Per subject microbiological cure rate | end of treatment and 7 to 14 days after the end of treatment
  The microbiological cure rate will be evaluated according to the microbiological identification results of the central laboratory
Per subject overall cure rate | end of treatment and 7 to 14 days after the end of treatment
  Evaluate the overall efficacy after a comprehensive consideration of the clinical results and the bacteriological results.
Safety evaluation | duration of trial
  Incidence and severity of AE and changes in safety parameters from baseline

CONTACTS AND LOCATIONS:
Locations (63):
- China (43):
  - Baotou Central Hospital, Baotou
  - Aerospace Center Hospital, Beijing
  - Affiliated Beijing Anzhen Hospital of Capital Medical University, Beijing
  - Affiliated Beijing Chaoyang Hospital of Capital Medical University, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing
  - Institute of Clinical Pharmacology, Peking University, Beijing
  - Peking University People's Hospital, Beijing
  - Changsha Central Hospital, Changsha
  - The Third Changsha Hotpital, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Daping Hospital, Chongqing
  - Guangxi Zhuang Autonomous Region People's Hospital, Guangxi
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Guilin Medical School Affiliated Hospital, Guilin
  - Hainan General Hospital, Haikou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - The First Hospital of Anhui Medical University, Hefei
  - The Affilated Hospital of Inner Mongolia Medical University, Hohhot
  - The First Hospital of Jilin University, Jilin
  - The Fourth Hospital of Jilin University, Jilin
  - Jinan Central Hospital, Jinan
  - The Second Hospital of Shandong University, Jinan
  - Gansu Provincial People's Hospital, Lanzhou
  - Jiangxi Provincial People's Hospital, Nanchang
  - Second Subsidiary Hospital of Nanchang Medical College, Nanchang
  - General Hospital of Nanjing Military Command, Nanjing
  - Institute of Antibiotics, Huashan Hospital, Fundan University, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shanghai East Hospital of Tongji University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - General Hospital of Shenyang Military, Shenyang
  - Shengjing Hospital, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The Second People's Hospital of Shenzhen, Shenzhen
  - General Hospital of Chengdu Military Region, Sichuan
  - West China Center of Medical Sciences of Sichuan University, Sichuan
  - First Hospital of Shanxi Medical University, Taiyuan
  - Wuxi People's Hospital, Wuxi
  - Tangdu Hospital, Xi'an
  - The First Affilated Hospital of Xiamen University, Xiamen
  - Northern Jiangsu People's Hospital, Yangzhou
  - The First Affiliated Hospital,College of Medicine,Zhejiang University, Zhejiang
- Taiwan (20):
  - Changhua Christian Hospital, Chang-hua
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - NTUH Hsin-Chu Branch, Hsinchu
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - Far Eastern Memorial Hospital, New Taipei City
  - MacKay Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University - Shuang Ho Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - NTUH Yun-Lin Branch, Yuli